CLINICAL TRIAL: NCT06568523
Title: A Multicenter Study to Evaluate the Diagnostic Performance of Computer-aided Polyp Size Classification of the MAGENTIQ-COLO During Real-time Colonoscopy
Brief Title: Study to Evaluate the Diagnostic Performance of of MAGENTIQ-COLO During Colonoscopy.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Magentiq Eye LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CL-0045
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Screening Colonoscopy; Surveillance Colonoscopy
Keywords: Colorectal Neoplasms; Intestinal Neoplasms; Digestive System Neoplasms; Screening Colonoscopy; Surveillance Colonoscopy; Automatic Polyp Detection
MeSH Terms: conditions — Colorectal Neoplasms; Intestinal Neoplasms; Digestive System Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Patients will undergo colonoscopy with the real-time use of the MAGENTIQ-COLO technology. (Other): Endoscopists will assess all colorectal polyps detected during colonoscopy with and without the MAGENTIQ-COLO.
  Interventions: Diagnostic Test: MAGENTIQ-COLO.

INTERVENTIONS:
Diagnostic Test: MAGENTIQ-COLO. — This is a diagnostic performance study; no randomization will be conducted. All subjects will undergo the same study procedures. The endoscopist performing the examinations cannot be blinded for the output of the investigational device in this study. Due to the nature of the intervention, it is not guaranteed that the patient is not awake during the procedure, therefore blinding for the patient is also not feasible.
  Other Names: Model: AI-DETECT-GI / AI-DETECT-GI-CU

SUMMARY:
This is an international, multicenter, study to evaluate the diagnostic performance of the CADx polyp sizing modality of the MAGENTIQ-COLO.

DETAILED DESCRIPTION:
Colonoscopy is the gold standard for the detection and removal of premalignant colorectal polyps. Recommended post-polypectomy surveillance intervals are primarily based on pathological diagnosis and polyp size. However, accurate estimation of polyp size remains challenging, potentially influencing post-polypectomy surveillance intervals. Inaccuracies in size estimation may lead to either unnecessary or prematurely scheduled surveillance colonoscopies when overestimating size or lead to an increased risk of post-colonoscopy colorectal cancer or advanced neoplasia when underestimating size. Furthermore, diminutive (1-5mm) polyps pose challenges due to their high incidence and frequent pathological assessment. Proposed strategies to reduce this burden, such as the European Society of Gastrointestinal Endoscopy (ESGE) 'resect-and-discard' strategy, are infrequently used as non-expert endoscopists often do not meet diagnostic thresholds when using standard visual inspection. The MAGENTIQ-COLO computer-aided diagnosis (CADx) system by Magentiq Eye LTD, Haifa, Israel, addresses these challenges by providing real-time polyp size estimation and polyp characterization. Additionally, this study evaluates the diagnostic accuracy of the MAGENTIQ-COLO CADx system in an average-risk screening and surveillance colonoscopy population.

The primary objective of the study is to assess the diagnostic performance of the endoscopist performing a MAGENTIQ-COLO CADx-assisted colonoscopy to classify polyps as diminutive (≤5mm) or non-diminutive (>5mm) compared to the size classification using open biopsy forceps, or polypectomy snares, of known diameter.

This will be measured by comparing the sensitivity and specificity between the two size classifications. Secondary objective include:

* To assess the diagnostic performance of the endoscopist performing a MAGENTIQ-COLO CADx-assisted colonoscopy to diagnose diminutive (rectosigmoid) colorectal polyps as neoplastic (adenoma or sessile serrated lesion (SSL)) with high-confidence compared to the pathology diagnosis. This will be measured by the sensitivity and specificity between the two diagnoses;
* To assess the diagnostic performance of the CADx system in measuring the size in millimeters and the size classification of colorectal polyps compared to the size measurement using open biopsy forceps, or polypectomy snare, of known diameter; this correlation will also be conducted for classifying polyps into diminutive (≤5mm), small (6-9mm), and advanced (≥10mm) size categories.

The sensitivity of the CADx-assisted optical diagnosis in classifying colorectal polyps as diminutive (≤5mm) or non-diminutive (>5mm) compared to the reference gold standard, which is the size classification of the colorectal polyp using open biopsy forceps, or polypectomy snare, of known diameter.

This is an international, multicenter, study to evaluate the diagnostic performance of the CADx polyp sizing modality of the MAGENTIQ-COLO. Study subjects who are already referred for screening or surveillance colonoscopy, will undergo colonoscopy with the real-time use of the MAGENTIQ-COLO technology. Endoscopists will assess all colorectal polyps detected during colonoscopy with and without the MAGENTIQ-COLO. Diagnostic performance of polyp size classification and optical diagnosis with and without MAGENTIQ-COLO is evaluated with reference to open biopsy forceps, or polypectomy snare of known diameter size classification, and pathology-based diagnosis, respectively. There is no formal study subject follow-up. Study procedures will be performed intraprocedural during the colonoscopy. Final pathological diagnosis will be recorded from the electronic health record.

The unit of analysis is the colorectal polyp rather than a study subject. The study is planned to include 396 colorectal polyps. Based on an expected detection rate of approximately 1.20 polyps per colonoscopy in the study population, we assume that enrollment of 330 subjects will be sufficient to meet the study objectives.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged ≥45 - ≤80 years old, who are scheduled for non-iFOBT screening or surveillance colonoscopy.

Exclusion Criteria:

1. In situ polyps with known histology detected in a previous colonoscopy.
2. No colorectal polyps detected during colonoscopy.
3. Known or suspected inflammatory bowel disease.
4. Polyposis syndrome (e.g., familial adenomatous polyposis, serrated polyposis).
5. Non-hereditary polyposis syndromes (e.g. Lynch syndrome).
6. History of chemotherapy or radiation therapy for colorectal lesions.
7. Pregnancy.
8. Has a referral for therapeutic procedure (i.e., endoscopic mucosal resection, intervention to stop a lower gastro-intestinal bleeding, etc.).
9. Inability to undergo polypectomy (e.g., incorrect continued use of anticoagulants, comorbidities) or patient refusal, as assessed by the endoscopist.
10. Inability to provide informed consent.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The sensitivity of the CADx-assisted optical diagnosis in classifying colorectal polyps as diminutive (≤5mm) or non-diminutive (>5mm) compared to the reference gold standard. | During the Colonoscopy Procedure
  The sensitivity of the CADx-assisted optical diagnosis in classifying colorectal polyps as diminutive (≤5mm) or non-diminutive (>5mm) compared to the reference gold standard, which is the size classification of the colorectal polyp using open biopsy forceps, or polypectomy snare, of known diameter.
  The diagnostic performance of the CADx-assisted optical diagnosis to correctly classify colorectal polyps as diminutive (≤5mm) or non-diminutive (>5mm) compared to size classification using open biopsy forceps, or polypectomy snare, of known diameter. This will be measured by the sensitivity and specificity of the CADx-assisted optical diagnosis compared to an expected minimum of 70% sensitivity and 70% specificity.

SECONDARY OUTCOMES:
CADx size measurement vs. open biopsy forceps | During the Colonoscopy Procedure
  The diagnostic performance of the optical diagnosis of the CADx system for correctly classifying colorectal polyps as diminutive (≤5mm) or non-diminutive (>5mm) compared to the size classification using open biopsy forceps, or polypectomy snare, of known diameter. This will be measured by the sensitivity, specificity, and accuracy of the CADx-assisted optical diagnosis.
  In addition, the correlation between the size measurement in millimeters by the CADx system and by using open biopsy forceps or polypectomy snare of known diameter will be calculated. This correlation will also be conducted for classifying polyps into diminutive (≤5mm), small (6-9mm), and advanced (≥10mm) size categories.
ESGE 'resect-and-discard' & 'leave-in-situ' | During the Colonoscopy Procedure
  The diagnostic performance of high-confidence CADx-assisted optical diagnosis to correctly identify diminutive colorectal polyps as neoplastic (adenoma or SSL). This will be measured by the sensitivity and specificity of the high-confidence CADx-assisted optical diagnosis compared to the ESGE 'resect-and-discard' strategy; an expected minimum of 80% sensitivity and 80% specificity. Additionally, for diminutive polyps located in the rectosigmoid, the diagnostic performance will be compared to the ESGE 'leave-in-situ' strategy, with an expected minimum sensitivity of 90% and specificity of 80% for neoplastic diagnosis

OTHER OUTCOMES:
ASGE PIVI-1 Post-polypectomy surveillance interval | During the Colonoscopy Procedure
  The ability of the CADx-assisted optical diagnosis to correctly assign post-polypectomy surveillance intervals. This will be measured by the agreement rate of high-confidence CADx-assisted optical diagnosis for polyps ≤5mm (cutoff based on the reference gold standard of this study) combined with the pathological diagnosis for polyps >5mm compared to the ASGE PIVI-1 criteria; an expected minimum of 90% agreement between assigning ASGE/US Multisociety Task Force on Colorectal Cancer (USMSTF) post-polypectomy surveillance intervals
ASGE PIVI-2 NPV of neoplastic rectosigmoid polyps | During the Colonoscopy Procedure
  The diagnostic performance of CADx-assisted optical diagnosis to correctly identify diminutive polyps in the rectosigmoid as neoplastic. This will be measured by the negative predictive value (NPV) of the high-confidence CADx-assisted optical diagnosis compared to the ASGE PIVI-2 criteria; an expected minimum of 90% NPV
Rate of high-confidence diagnoses | During the Colonoscopy Procedure
  The rate of high-confidence neoplastic diagnoses (size and optical diagnosis) of diminutive colorectal polyps between standard visual inspection, the CADx system diagnosis, and CADx-assisted optical diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Siersema, MD, Ph.D., Principal Investigator — Erasmus Medical Center
Locations (5):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Erlanger Health System, Chattanooga, Tennessee
- Israel (2):
  - Assuta, Haifa, Select State
  - Hadassah Medical Organization, Jerusalem
- Erasmus Medical Center, Rotterdam, Netherlands